CLINICAL TRIAL: NCT00345345
Title: Treatment of T-Large Granular Lymphocyte (T-LGL) Lymphoproliferative Disorders With Alemtuzumab (Campath)
Brief Title: Alemtuzumab (Campath) to Treat T-Large Granular Lymphocyte Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060190; 06-H-0190; NCT00365066 (obsolete NCT alias)
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-03

CONDITIONS: T-LGL Lymphoproliferative Disorders
Keywords: Neutropenia; Monoclonal Antibody Therapy; Anti-CD52; T-LGL Leukemia; LGL Leukemia; Leukemia
MeSH Terms: conditions — Neutropenia; Leukemia, Large Granular Lymphocytic; Leukemia | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alemtuzumab in patients with T cell large granular lymphocytic leukemia (T-LGL) (Experimental): Alemtuzumab (Campath) will be administered at 10 mg/dose IV for 10 days as an infusion over 2 hours.
  Interventions: Biological: Alemtuzumab (Campath)

INTERVENTIONS:
Biological: Alemtuzumab (Campath) — Alemtuzumab (Campath) will be administered at 10 mg/dose IV for 10 days as an infusion over 2 hours.

SUMMARY:
This study will examine the use of alemtuzumab (Campath) in patients with T cell large granular lymphocytic leukemia (T-LGL). Patients with T-LGL often have reduced white blood cells, red blood cells and platelets, and increased numbers of abnormal cells called large granular lymphocytes (LGLs). Patients may have recurrent infections, anemia, or abnormal bleeding. Campath destroys specific parts of the abnormal LGLs, which interfere with the production of normal blood cells. This study will determine whether Campath can increase blood counts and reduce the number of abnormal LGLs in patients and will examine the side effects of the drug.

Patients 18 to 85 years of age with T-LGL leukemia may be eligible for this study. Participants undergo the following procedures:

Before starting Campath treatment

* Medical history and physical examination, blood tests, electrocardiogram (ECG).
* Echocardiogram (heart ultrasound) and 24-hour Holter monitoring (continuous ECG recording).
* Bone marrow biopsy: About a tablespoon of bone marrow is withdrawn through a needle inserted into the hipbone. The procedure is done using local anesthetic.
* Placement of central line, if needed: An intravenous line (tube) is placed into a major vein in the chest. It can stay in the body and be used for the entire treatment period. The line is used to give chemotherapy or other medications, including antibiotics and blood transfusions, and to collect blood samples. The line is usually placed under local anesthesia in the radiology department or the operating room.
* Apheresis: A catheter (plastic tube) is placed in a vein in each arm. Blood is drawn from one vein and run through a cell-separating machine, where the white blood cells are collected and saved. The remaining blood is transfused back to the patients through the vein in the other arm.

During Campath treatment

* Campath therapy: After a small test dose, patients receive10 daily infusions of Campath, each of which lasts about 2 hours. The first few infusions are given at the NIH Clinical Center so that the patient can be monitored closely.
* Induction therapy: Aerosolized pentamadine, valacyclovir and other medicines are given to protect against or treat various infections that commonly affect patients with suppressed immune systems.
* Whole blood or platelet transfusions, if needed, and injections of growth factors, if needed.
* Blood tests and check of vital signs (temperature, pulse, blood pressure) every day during treatment. Echocardiogram and 24-hour Holter monitor after the last dose of Campath.

Follow-up evaluations after Campath treatment ends

* Blood tests at home or at NIH (weekly for the first 3 months, then every other week until 6 months, then annually for 5 years
* Echocardiogram at NIH (at 3 months only)
* Bone marrow biopsy at NIH (at 6 and 12 months, then as clinically indicated)
* One repeat apheresis collection for laboratory studies.

DETAILED DESCRIPTION:
T Cell Large Granular Lymphocyte (T-LGL) lymphoproliferative disorders are a heterogeneous group of uncommon diseases which may involve a monoclonal or oligoclonal T cell population, which bear characteristic surface markers corresponding to activated cytotoxic (CD3+, CD8+) lymphocytes. They are often associated with quite severe neutropenia, anemia, and thrombocytopenia, which may be life-threatening. There is some evidence that the abnormal cytotoxic lymphocyte population may cause the cytopenias by suppressing hematopoiesis, although the mechanism is unclear. Immunosuppressive therapy has been shown to improve the cytopenias of T-LGL leukemia, however the long-term use of the commonly used agents often lead to significant toxicity in the older patients which are affected by this disease.

Alemtuzumab (Campath[R]) is currently approved as second line agent in patients with chronic lymphocytic leukemia (CLL) and has been used successfully in the treatment of certain autoimmune disorders. In the Hematology Branch, Campath is currently being investigated in two bone marrow failure syndromes: aplastic anemia and myelodysplasia. Cytopenia(s) is an important characteristic of patients with T-LGL leukemia, often being the indication for immunosuppressive therapy. Our preliminary experience with Campath indicates that it is well tolerated, among the elderly patients.

Therefore, we propose this pilot, Phase II, single agent, study which will evaluate the efficacy and safety of alemtuzumab (Campath[R]), an immunosuppressive drug, in subjects with T-LGL leukemia. Commercially available Alemtuzumab (Campath[R]) will be administered off label at 10 mg per day by intravenous infusion for 10 days total. Subjects who do not show a response to initial Campath or relapse may receive a second cycle of drug after the 3-month time point.

The primary end point of the study is the response rate at three months, defined as improvement in cytopenia(s). Secondary endpoints will include relapse-free survival, response at 6 months, life threatening toxicity, reduction in the number of abnormal T-LGL clone, response to second cycle of Campath, and overall survival.

ELIGIBILITY:
* INCLUSION CRITERIA:

Clinical history supportive of the diagnosis of T-LGL leukemia (i.e. a history of cytopenias with peripheral blood morphologic evidence of LGLs)

Immunophenotypic studies of peripheral blood showing an increased population of T-LGLs (suggested by staining with CD3+, CD8+ and CD16+ or CD57+) or gammadelta T cells

Restricted or clonal rearrangement of the T-cell receptor by PCR AND one or more of the following:

Severe neutropenia (less than 500 neutrophils/microliter); OR

Severe thrombocytopenia (less than 20,000 platelets/microliter), or moderate thrombocytopenia (less than 50,000 platelets/microliter) with active bleeding; OR

Symptomatic anemia with a hemoglobin less than 9 g/dL or red blood cell transfusion requirement of greater than 2 units/month for two months prior to initiation of Campath

Ages 18-85 (both inclusive)

EXCLUSION CRITERIA:

A reactive LGL lymphocytosis to a viral infection

Serologic evidence of HIV infection

Infection not adequately responding to appropriate therapy

Previous immunosuppressive therapy with alemtuzumab

History of carcinoma that is not considered cured (excluding non-melanoma skin carcinoma)

Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the subject's ability to tolerate protocol therapy or that death within 7-10 days is likely

Current pregnancy or unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential

Not able to understand the investigational nature of the study or give informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-10-17 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan F Cordes, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] McKenna RW, Parkin J, Kersey JH, Gajl-Peczalska KJ, Peterson L, Brunning RD. Chronic lymphoproliferative disorder with unusual clinical, morphologic, ultrastructural and membrane surface marker characteristics. Am J Med. 1977 Apr;62(4):588-96. doi: 10.1016/0002-9343(77)90422-3. PMID 192076
- [Background] Loughran TP Jr. Clonal diseases of large granular lymphocytes. Blood. 1993 Jul 1;82(1):1-14. PMID 8324214
- [Background] Semenzato G, Zambello R, Starkebaum G, Oshimi K, Loughran TP Jr. The lymphoproliferative disease of granular lymphocytes: updated criteria for diagnosis. Blood. 1997 Jan 1;89(1):256-60. PMID 8978299
- [Derived] Dumitriu B, Ito S, Feng X, Stephens N, Yunce M, Kajigaya S, Melenhorst JJ, Rios O, Scheinberg P, Chinian F, Keyvanfar K, Battiwalla M, Wu CO, Maric I, Xi L, Raffeld M, Muranski P, Townsley DM, Young NS, Barrett AJ, Scheinberg P. Alemtuzumab in T-cell large granular lymphocytic leukaemia: interim results from a single-arm, open-label, phase 2 study. Lancet Haematol. 2016 Jan;3(1):e22-9. doi: 10.1016/S2352-3026(15)00227-6. Epub 2015 Dec 17. PMID 26765645
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-H-0190.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Alemtuzumab in Patients With T Cell Large Granular Lymphocytic Leukemia (T-LGL): 10 mg Alemtuzumab (Campath®; Genzyme) was administered intravenously daily for 10 days, after a 1 mg intravenous test dose.
Period: Overall Study
Arm/Group | Alemtuzumab in Patients With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Started | 29
Completed | 27
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab in Patients With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hematological Response After Three Months of Alemtuzumab
Description: The primary endpoint was hematologic response at three months after treatment. A complete response (CR) was defined as normalization of all affected lineages, and a partial response (PR) was defined in neutropenic subjects as 100% increase in the ANC to >500/µL, and in those with anemia, any increase in hemoglobin of 2 g/dL or more observed in at least two serial measurements 1 week apart and sustained for one month or more without exogenous growth factors support or transfusions.
Time Frame: 3 months
Population: The analyses included only those subjects who were given Alemtuzumab. Analysis was by intention to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab in Patients With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 29
Participants | 15

2. Secondary Outcome: Number of Participants That Are Red Blood Cell and/or Platelet Transfusion-Independent
Description: Number of participants that are red blood cell and/or platelet Transfusion-Independent following Alemtuzumab
Time Frame: 3 months
Population: Analysis was by intention to treat. One participant not evaluable, died prior to 3 months.
Measure: Count of Participants; unit: Participants
Groups:
- Alemtuzumab in Participants With T Cell Large Granular Lymphocytic Leukemia (T-LGL): 10 mg Alemtuzumab (Campath®; Genzyme) was administered at 10 mg/dose intravenously daily for 10 days over 2 hours, after a 1 mg intravenous test dose.
Arm/Group | Alemtuzumab in Participants With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 28
Participants
  Both red blood cell and platelet transfusion-independent | 16
  Either red blood cell or platelet transfusion-dependent | 12

3. Secondary Outcome: Participants Overall Survival After Alemtuzumab Infusion
Description: Participants overall survival after Alemtuzumab infusion for cell large granular lymphocytic leukemia (T-LGL) at month 3.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab in Participants With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 29
Participants
  Alive | 28
  Deceased | 1

4. Secondary Outcome: Number of Participants That Experienced a Life-Threatening Toxicity
Description: Number of participants that experienced a Life-Threatening Toxicity (grade >/= 4) as defined by Common toxicity Criteria (CTC) version 2.0. The CTC 2.0 is a set of criteria for the standardized classification of adverse effects. Adverse events are graded accordingly: 0 = No adverse event or within normal limits 1 = Mild adverse event 2 = Moderate adverse event 3 = Severe and undesirable adverse event 4 = Life-threatening or disabling adverse event 5 = Death related to adverse event
Time Frame: 12 months
Population: Analysis was by intention to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab in Patients With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 29
Participants
  Lymphocyte count decreased | 13
  White blood cell decreased | 3
  Platelet count decreased | 2
  Neutrophil count decreased | 1
  Monocytes count decreased | 1

5. Secondary Outcome: Number of Participants That Are Relapse-free Survival Following Campath Infusion.
Description: Number of participants that are Relapse-free survival following Campath infusion. Relapse is defined as a fall in peripheral blood counts to 50% the values obtained during the response period.
Time Frame: Month 12
Population: 10 participants were not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab in Participants With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 19
Participants | 10

6. Secondary Outcome: Number of Participants With Molecular Response to Campath
Description: Number of Participants with Molecular Response to Campath. Molecular Response to Campath is defined as disappearance of the clonal population of T-LGL
Time Frame: Up to Month 12
Population: Participants who completed molecular testing
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab in Participants With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 21
Participants | 14

7. Secondary Outcome: Participant Response at 6 Months
Description: Participant response at 6 months following Alemtuzumab. A complete response (CR) was defined as normalization of all affected lineages, and a partial response (PR) was defined in neutropenic subjects as 100% increase in the ANC to >500/µL, and in those with anemia, any increase in hemoglobin of 2 g/dL or more observed in at least two serial measurements 1 week apart and sustained for one month or more without exogenous growth factors support or transfusions.
Time Frame: 6 months
Population: 5 participants were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab in Participants With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 24
Participants
  Complete Response | 10
  No Response | 5
  Disease Relapse | 4
  Partial Response | 5

8. Secondary Outcome: Participants Response to a Second Cycle of Campath
Description: Participants Response to a second cycle of Campath. A complete response (CR) was defined as normalization of all affected lineages, and a partial response (PR) was defined in neutropenic subjects as 100% increase in the ANC to >500/µL, and in those with anemia, any increase in hemoglobin of 2 g/dL or more observed in at least two serial measurements 1 week apart and sustained for one month or more without exogenous growth factors support or transfusions.
Time Frame: 12 months
Population: Participants that received a second cycle of Campath
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab in Participants With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 8
Participants
  No response | 5
  Relapsed | 3
  Complete Response | 0
  Partial Response | 0

9. Secondary Outcome: Number of Participants With Clone Size Improvements
Description: Number of participants with clone size improvements following Alu
Time Frame: Up to 6 months
Population: 3 participants were not evaluable as no data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab in Participants With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
Number analyzed (Participants) | 26
Participants
  Deceased in clone size | 20
  No deceased in clone size | 6

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Alemtuzumab in Patients With T Cell Large Granular Lymphocytic Leukemia (T-LGL)
All-Cause Mortality (participants affected / at risk) | 8/29
Serious Adverse Events (participants affected / at risk) | 13/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab in Patients With T Cell Large Granular Lymphocytic Leukemia (T-LGL) (N=29)
Acquired dysfibrinogenaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Atrial fibrillation (Cardiac disorders) | 1
Autoimmune colitis (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Injection site infection (General disorders) | 1
Bacterial infection (Infections and infestations) | 2
Clostridium difficile infection (Infections and infestations) | 2
Mycobacterial infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Hemoglobin decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Respiratory failure (Metabolism and nutrition disorders) | 1
Aortic aneurysm repair (Surgical and medical procedures) | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab in Patients With T Cell Large Granular Lymphocytic Leukemia (T-LGL) (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Petechiae (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Chest discomfort (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 2
Dizziness (Cardiac disorders) | 5
Dizziness postural (Cardiac disorders) | 1
Dyspnea (Cardiac disorders) | 5
Dyspnea exertional (Cardiac disorders) | 2
Fluid overload (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Peripheral swelling (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Ear infection (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Blepharitis (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Ophthalmic herpes simplex (Eye disorders) | 1
Photopsia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Diverticulitis (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 2
Eructation (Gastrointestinal disorders) | 1
Gastroenteritis viral (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Oral herpes (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Oropharyngeal candidiasis (Gastrointestinal disorders) | 1
Oropharyngeal pain (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 3
Chills (General disorders) | 15
Crepitations (General disorders) | 1
Decreased appetite (General disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 7
Feeling hot (General disorders) | 1
Gait disturbance (General disorders) | 1
Hyperhidrosis (General disorders) | 2
Infusion related reaction (General disorders) | 12
Injection site hemorrhage (General disorders) | 3
Injection site pain (General disorders) | 1
Malaise (General disorders) | 1
Night sweats (General disorders) | 2
Oedema (General disorders) | 3
Peripheral coldness (General disorders) | 1
Pyrexia (General disorders) | 15
Swelling (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Urticaria (Immune system disorders) | 1
Bacteremia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Iron overload (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood electrolytes decreased (Investigations) | 1
Blood fibrinogen increased (Investigations) | 1
Blood glucose increased (Investigations) | 2
Blood iron decreased (Investigations) | 1
Blood pressure decreased (Investigations) | 2
Blood pressure increased (Investigations) | 5
Blood thyroid stimulating hormone increased (Investigations) | 3
Ejection fraction decreased (Investigations) | 1
Heart rate decreased (Investigations) | 1
Heart rate increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 5
Liver function test abnormal (Investigations) | 2
Lymphocyte count decreased (Investigations) | 25
Monocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Oxygen saturation decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Prothrombin time prolonged (Investigations) | 3
Transaminases increased (Investigations) | 1
Troponin increased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell counts decreased (Investigations) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Restless legs syndrome (Musculoskeletal and connective tissue disorders) | 1
Sciatica (Musculoskeletal and connective tissue disorders) | 1
Confusional state (Nervous system disorders) | 1
Headache (Nervous system disorders) | 9
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 4
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 5
Thrombophlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT00345345/Prot_SAP_000.pdf